CLINICAL TRIAL: NCT02304991
Title: Peanut Sublingual Immunotherapy Induction of Clinical Tolerance of Newly Diagnosed Peanut Allergic 12 to 48 Month Old Children
Brief Title: FARE Peanut SLIT and Early Tolerance Induction
Acronym: FARE/SLIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Food Allergy Research & Education (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0648; R01AT004435-07 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-01

CONDITIONS: Peanut Hypersensitivity; Food Allergy; Food Hypersensitivity; Peanut Allergy
Keywords: Peanut; Food Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut (liquid peanut extract) SLIT (Experimental): After the entry DBPCFC, subjects will be randomized 1:1 to active or placebo drug product. Subjects randomized to peanut SLIT therapy will dose for 36 months and undergo a second DBPCFC. The subjects will stop dosing for three months and repeat a DBPCFC at 39 months.
  Interventions: Drug: Liquid Peanut Extract
- Placebo Glycerin SLIT (Placebo Comparator): After the entry DBPCFC, subjects will be randomized 1:1 to active or placebo drug product. Subjects randomized to placebo glycerin SLIT will dose for 36 months and undergo a second DBPCFC. The subjects will stop dosing for three months and repeat a DBPCFC at 39 months.
  Interventions: Drug: Placebo Glycerin SLIT

INTERVENTIONS:
Drug: Liquid Peanut Extract — 5000mcg/ml peanut protein
  Other Names: SLIT
  Arms: Peanut (liquid peanut extract) SLIT
Drug: Placebo Glycerin SLIT — pure glycerinated saline solution with caramel coloring to match color
  Other Names: SLIT
  Arms: Placebo Glycerin SLIT

SUMMARY:
Primary Objective: To determine if 36 months of peanut SLIT as an early intervention in subjects ages 1 to 4 years induces clinical desensitization. The primary outcome of this objective will be a statistically significant difference in challenge scores between the treatment group versus the placebo group during DBPCFC (Double blind placebo controlled food challenge) performed after 36 months of peanut SLIT (desensitization). Challenge scores are measured by the amount of peanut protein participants are able to ingest successfully without symptoms of an allergic reaction. [Time Frame: Baseline, 36 months]

Secondary Objectives:

A secondary outcome of this objective will be a statistically significant difference in the challenge score of the treatment group versus the placebo group during the DBPCFC performed 3 months after discontinuing therapy (tolerance).

To examine the change in immune parameters associated with peanut SLIT and the development of clinical tolerance. Through this objective, the investigators will seek to understand the molecular processes by which SLIT affects the immune system through evaluation of immune mechanisms in relationship to clinical findings of desensitization and tolerance. The investigators will delineate the impact of peanut SLIT on the subsequent cellular and humoral responses to peanut protein.

[Time Frame: Baseline, 39 months]

DETAILED DESCRIPTION:
Peanut allergy is one of the most common food allergies; most children develop this allergy early in life, do not outgrow it and are at risk for severe and life-ending anaphylactic reactions. There is a critical need for a proactive treatment for peanut allergy and the investigators along with others are developing specific types of immunotherapy that will act as disease-modifying therapies.

This SLIT study is a randomized, blinded, placebo-controlled study. The primary outcome of this objective will be a statistically significant difference in challenge scores between the treatment group versus the placebo group during DBPCFC performed after 36 months of peanut SLIT (desensitization). A secondary outcome of this objective will be a statistically significant difference in the challenge score of the treatment group versus the placebo group during the DBPCFC performed 3 months after discontinuing therapy (tolerance).

Upon enrollment into the study, all subjects will undergo a qualifying entry DBPCFC with peanut protein to confirm the diagnosis of peanut allergy and establish a baseline threshold level. Following a positive DBPCFC, each subject will be randomized 1:1 to receive peanut SLIT therapy versus placebo for a duration of 36 months. DBPCFC will be repeated for both active and placebo subjects at 36 months to assess desensitization and at 39 months to assess tolerance.

Outcome variables of interest include peanut specific IgE, IgG, and IgG4, basophil activation, mast cell responses through skin prick testing, and specific T-cell cytokine responses and T regulatory cell (TReg) activation.

COVID-19 SAFETY MEASURES- Reflected in Protocol V4.0- April 2020

In March of 2020, State and National emergencies were declared over the global pandemic coronavirus COVID-19.

As such, any 36 month Desensitization DBPCFC will be postponed while the safety measures surrounding COVID-19 are in place. Subjects who choose to remain in the study will continue on study drug at the maintenance dose level beyond the originally planned 36 months until such time that the Desensitization DBPCFC is conducted.

Subjects who are scheduled to undergo the 39 month Tolerance DBPCFC while the COVID-19 safety measures are in place will have their DBPCFC cancelled. Additional time off of study drug therapy would potentially increase the risk of allergic reaction during the DBPCFC and would not be acceptable.

For subjects whose Desensitization DBPCFC is postponed, a followup visit to review safety and subject dosing diaries would be conducted. This visit would be conducted remotely by telephone. Additional study drug would be sent direct-to-patient as necessary to continue on maintenance dosing. Lab sample collection and mechanistic studies would be deferred and be completed at the time that the Desensitization DBPCFC is completed. The Tolerance DBPCFC would be completed 3 months after the Desensitization DBPCFC is completed.

For subjects whose Tolerance DBPCFC is canceled, an exit visit would be conducted to review safety. The subject would be unblinded to treatment allocation and end of study instructions would be reviewed with the subject.

As the situation is changing daily, we are unable to provide a time frame for extension. We hope to limit the number of subjects who will need to utilize this option and preserve the endpoint data parameters. Previous SLIT studies have not shown any additional risk with peanut SLIT dosing beyond 3 years up to a total of 5 years of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from participant's parent/guardian.
* Age 12-48 months of either sex, any race, any ethnicity.
* A peanut allergy diagnosis with a convincing clinical history of peanut allergy and a serum peanut-specific IgE [UniCAP] > 0.35 kUA/L AND a positive skin prick test to peanut (>3 mm than the negative control) OR are sensitized to peanut (based on a serum IgE [UniCAP] to peanut of > 5 kUA/L) AND a positive skin prick test to peanut (> 3 mm than the negative control) and no known history of ingestion of peanut.
* A positive DBPCFC to 1000 mg of peanut at enrollment.

Exclusion Criteria:

* History of severe anaphylaxis to peanut, defined as hypoxia, hypotension, or neurologic compromise (cyanosis or peripheral capillary oxygen saturation (SpO2) < 92% at any stage, hypotension, confusion, collapse or loss of consciousness).
* Participation in any interventional study for the treatment of food allergy in the past 6 months.
* Known oat, wheat, or glycerin allergy.
* Eosinophilic or other inflammatory (e.g. celiac) gastrointestinal disease.
* Severe asthma (2007 NHLBI Criteria Steps 5 or 6 - Appendix 2).
* Inability to discontinue antihistamines for skin testing and DBPCFCs.
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immunomodulator therapy (not including corticosteroids) or biologic therapy within the past year.
* Use of beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers.
* Significant medical condition (e.g., liver, kidney, gastrointestinal, cardiovascular, hematologic, or pulmonary disease) which would make the subject unsuitable for induction of food reactions.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peanut (Liquid Peanut Extract) SLIT: After the Double-Blind, Placebo-Controlled Food Challenge (DBPCFC), subjects randomized 1:1 to active or placebo drug product. Subjects randomized to peanut SLIT therapy will dose for 36 months and undergo a second DBPCFC. The subjects will stop dosing for three months and repeat a DBPCFC at 39 months.
  Liquid Peanut Extract: 5000mcg/ml peanut protein
- Placebo Glycerin SLIT: After the Double-Blind, Placebo-Controlled Food Challenge (DBPCFC), subjects randomized 1:1 to active or placebo drug product. Subjects randomized to placebo glycerin SLIT will dose for 36 months and undergo a second DBPCFC. The subjects will stop dosing for three months and repeat a DBPCFC at 39 months.
  Placebo Glycerin SLIT: pure glycerinated saline solution with caramel coloring to match color
Period: Overall Study
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Started | 25 | 25
Completed | 18 | 15
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 2.2 [1.1 to 3.9] | 2.4 [1.0 to 4.0] | 2.2 [1.0 to 4.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 21 | 23 | 44
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
Peanut-Specific IgE [Mean (Full Range); unit: kUA/L] | 28.1 [0.3 to 180.0] | 37.8 [0.8 to 113.0] | 32.2 [0.3 to 180.0]
Peanut Skin Prick Test Wheal Size [Mean (Full Range); unit: mm] | 11.0 [4.0 to 20.5] | 11.2 [5.5 to 24.5] | 11.1 [4.0 to 24.5]

OUTCOME MEASURES:

1. Primary Outcome: Desensitization After 36 Months of Peanut SLIT or Placebo SLIT
Description: The primary outcome of this study will be a statistically significant difference in the challenge score of the treatment group versus the placebo group during DBPCFC after 36 months of peanut SLIT (desensitization).
  DBPCFC Challenge Score scale:
  Minimum score = 0; Maximum score = 7 Larger challenge score equals more successful desensitization. 0mg = 0; 3mg = 1; 13mg = 2; 43mg = 3; 143mg = 4; 443mg = 5; 1443mg = 6; and 4443mg = 7.
Time Frame: 36 months
Population: Intent to treat; participants not completing the DBPCFC considered to have challenge score of zero
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Number analyzed (Participants) | 25 | 25
score on a scale | 4.9 [3.7 to 6.2] | 2.5 [1.6 to 3.3]
Statistical Analysis 1: Comparison: Peanut (Liquid Peanut Extract) SLIT vs Placebo Glycerin SLIT; Intent to treat; participants not completing the DBPCFC considered to have challenge score of zero; Test type: Superiority; p = 0.002, t-test, 2 sided

2. Secondary Outcome: Tolerance 3 Months After Discontinuing Peanut SLIT or Placebo SLIT
Description: A secondary outcome of this study will be a statistically significant difference in the challenge score of the treatment group versus the placebo group during the DBPCFC performed 3 months after discontinuing therapy (tolerance).
  DBPCFC Challenge Score scale:
  Minimum score = 0; Maximum score = 7 Larger challenge score equals more successful desensitization. 0mg = 0; 3mg = 1; 13mg = 2; 43mg = 3; 143mg = 4; 443mg = 5; 1443mg = 6; and 4443mg = 7.
Time Frame: 39 months
Population: Intent to treat; participants not completing the DBPCFC considered to have challenge score of zero
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Number analyzed (Participants) | 25 | 25
score on a scale | 4.0 [2.6 to 5.4] | 1.0 [0.0 to 1.9]
Statistical Analysis 1: Comparison: Peanut (Liquid Peanut Extract) SLIT vs Placebo Glycerin SLIT; Intent to treat; participants not completing the DBPCFC considered to have challenge score of zero; Test type: Superiority; p = 0.0005, t-test, 2 sided

3. Secondary Outcome: Change in Immune Parameters With Peanut SLIT Versus Placebo SLIT (Peanut-specific IgE)
Description: The change in immune parameters over time associated with the induction of clinical desensitization compared to the failure to achieve clinical desensitization.
  Peanut-specific IgE measured at baseline and at completion of peanut SLIT (36 months). Change in IgE reported in kUA/L.
Time Frame: 0 months to 36 months
Population: Per protocol analysis of patients with available samples.
Measure: Mean (95% Confidence Interval); unit: kUA/L of peanut-specific IgE
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Number analyzed (Participants) | 17 | 12
kUA/L of peanut-specific IgE | -19.4 [-39.6 to 0.8] | 65.2 [-6.2 to 136.5]
Statistical Analysis 1: Comparison: Peanut (Liquid Peanut Extract) SLIT vs Placebo Glycerin SLIT; Test type: Superiority; p = 0.007, t-test, 2 sided

4. Secondary Outcome: Change in Immune Parameters With Peanut SLIT Versus Placebo SLIT (Peanut-specific IgG4)
Description: The change in immune parameters over time associated with the induction of clinical desensitization compared to the failure to achieve clinical desensitization.
  Peanut-specific IgG4 measured at baseline and at completion of peanut SLIT (36 months). Change in IgG4 reported in mg/L.
Time Frame: 0 months to 36 months
Population: Per protocol analysis of patients with available samples.
Measure: Mean (95% Confidence Interval); unit: mg/L of peanut-specific IgG4
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Number analyzed (Participants) | 17 | 11
mg/L of peanut-specific IgG4 | 3.9 [1.7 to 6.1] | -0.2 [-1.8 to 1.5]
Statistical Analysis 1: Comparison: Peanut (Liquid Peanut Extract) SLIT vs Placebo Glycerin SLIT; Per protocol analysis of patients with available samples; Test type: Superiority; p = 0.01, t-test, 2 sided

5. Secondary Outcome: Change in Immune Parameters With Peanut SLIT Versus Placebo SLIT (Peanut Skin Prick Test)
Description: The change in immune parameters over time associated with the induction of clinical desensitization compared to the failure to achieve clinical desensitization.
  Peanut-skin prick test measured at baseline and at completion of peanut SLIT (36 months). Change in skin prick test reported in mm wheal diameter.
Time Frame: 0 months to 36 months
Population: Per protocol analysis of patients with available samples.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Number analyzed (Participants) | 20 | 18
mm | -7.7 [-9.8 to -5.6] | 1.8 [-1.4 to 4.9]
Statistical Analysis 1: Comparison: Peanut (Liquid Peanut Extract) SLIT vs Placebo Glycerin SLIT; Per protocol analysis of patients with available samples; Test type: Superiority; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events With Peanut SLIT Versus Placebo SLIT
Description: Incidence of all serious adverse events from initial enrollment through the end of the 3 month avoidance period reported as the number of participants experiencing a serious adverse event.
Time Frame: 39 months
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
Number analyzed (Participants) | 25 | 25
Participants | 0 | 1
Statistical Analysis 1: Comparison: Peanut (Liquid Peanut Extract) SLIT vs Placebo Glycerin SLIT; Test type: Superiority; p = 0.3, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning with completion of the qualifying DBPCFC and enrollment in the study through the completion of the tolerance DBPCFC at the 39 month study time point.
Arm/Group | Peanut (Liquid Peanut Extract) SLIT | Placebo Glycerin SLIT
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 24/25 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peanut (Liquid Peanut Extract) SLIT (N=25) | Placebo Glycerin SLIT (N=25)
Acute Lymphoblastic Leukemia (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peanut (Liquid Peanut Extract) SLIT (N=25) | Placebo Glycerin SLIT (N=25)
Skin (Skin and subcutaneous tissue disorders) | 20 | 17
Gastrointestinal (Gastrointestinal disorders) | 11 | 8
Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Lower respiratory (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Oropharyngeal itch (Skin and subcutaneous tissue disorders) | 20 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02304991/Prot_SAP_000.pdf